CLINICAL TRIAL: NCT05112848
Title: A Phase 2, Randomized, Observer-Blinded Study to Evaluate the Safety and Immunogenicity of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine (SARS-CoV-2 rS) With Matrix-M™ Adjuvant in People Living With HIV
Brief Title: A Study to Evaluate Safety and Immunogenicity of a COVID-19 Vaccine in People Living With HIV at Risk for SARS-CoV-2 (COVID-19)
Acronym: COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019nCoV-505
Record Dates: First submitted 2021-10-25; First posted 2021-11-09 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV-2 Infection
Keywords: Coronavirus disease 2019 (COVID-19); HIV
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 PLWH (Experimental): Two doses of 5μg monovalent prototype vaccine+50µg Matrix-M adjuvant, given on Day 0 and Day 21.
  Alternating IM (deltoid) injection of placebo (0.5mL) given on Day 70.
  Interventions: Biological: NVX-CoV2373
- Group 2 PLWH (Experimental): Three doses of 5μg monovalent prototype vaccine+50µg Matrix-M adjuvant, given on Day 0, Day 21, and Day 70.
  Interventions: Biological: NVX-CoV2373
- Group 3 PLWH (Experimental): Two doses of 5μg monovalent prototype vaccine+50µg Matrix-M adjuvant, given on Day 0 and Day 70.
  Alternating IM (deltoid) injection of placebo (0.5mL) given on Day 21.
  Interventions: Biological: NVX-CoV2373
- Group 4 HIV-Negative Participants (Experimental): 2 doses of 5μg monovalent prototype vaccine+50µg Matrix-M adjuvant, given on Day 0 and Day 21.
  Alternating IM (deltoid) injection of placebo (0.5mL) given on Day 70.
  Interventions: Biological: NVX-CoV2373
- Group 5 HIV-Negative Participants (Experimental): Two doses of 5μg monovalent prototype vaccine+50µg Matrix-M adjuvant, given on Day 0 and Day 70.
  Alternating IM (deltoid) injection of placebo (0.5mL) given on Day 21.
  Interventions: Biological: NVX-CoV2373

INTERVENTIONS:
Biological: NVX-CoV2373 — Alternating intramuscular (IM) (deltoid) injections of monovalent prototype vaccine premixed with Matrix-M™ adjuvant (0.5 mL) given either as
  2 doses (one on Day 0 and one on Day 21 or Day 70) and an injection of placebo (0.5mL) on Day 21 or Day 70, or 3 doses (Day 0, Day 21, and Day 70).
  Other Names: Monovalent SARS-CoV-2 rS vaccine premixed with Matrix-M adjuvant

SUMMARY:
This is a Phase 2, randomized, observer-blinded study evaluating the safety and immunogenicity of SARS-CoV-2 with Matrix-M™ Adjuvant in people living with human immunodeficiency virus (HIV) (PLWH) and HIV- negative adults, seronegative to SARS-CoV-2 at baseline.

DETAILED DESCRIPTION:
The investigational product will be a monovalent Serum Institute of India (SII) SARS CoV-2 vaccine at a dose of 5 µg antigen adjuvanted with 50 µg Matrix-M (referred hereafter as NVX-CoV2373).

Approximately 270 PLWH, 18 to 65 years of age inclusive, will be enrolled into 3 groups and stratified at presentation based on the level of control of HIV infection. All PLWH will be baseline seronegative (for SARS-CoV-2) and have not received any authorized SARS-CoV-2 vaccines. PLWH will be randomly assigned 1:1:1 to receive NVX-CoV2373 in either a two dose regimen on Days 0 and 21 or Days 0 and 70 or a three-dose regimen on Days 0, 21, and 70. Randomization of PLWH will be stratified by level of control of HIV infection to distribute well controlled and less well controlled participants approximately evenly among the 3 PLWH treatment groups. Approximately 90 HIV negative participants, 18 to 65 years of age inclusive, will be randomly assigned 1:1 to receive NVX-CoV2373 in a two dose regimen on Days 0 and 21 or Days 0 and 70. All HIV negative participants will be baseline seronegative (for SARS-CoV-2) and have not received any authorized SARS-CoV-2 vaccines. Placebo (normal saline solution) will be administered to participants who receive a two-dose regimen of NVX-CoV2373 to maintain overall blinding.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 65 years of age, inclusive, at screening.
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from at least 28 days prior to enrollment and through the end of the study.

   1. Condoms (male or female) with spermicide (if acceptable in-country)
   2. Diaphragm with spermicide
   3. Cervical cap with spermicide
   4. Intrauterine device
   5. Oral or patch contraceptives
   6. Norplant®, Depo-Provera®, or other in-country regulatory approved contraceptive method that is designed to protect against pregnancy.
   7. Abstinence as a form of contraception is acceptable if in line with the participant's lifestyle.
4. Vital signs must be within medically acceptable ranges prior to the first vaccination
5. Agree to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study.

   For well-controlled PLWH
6. PLWH with a cluster of differentiation 4 (CD4) + T-cell count of ≥ 350 cells/μL at screening or viral load of ≤ 1,000 copies/mL.
7. PLWH being managed on a stable/unchanged antiretroviral therapy (ART) regimen for at least 2 months prior to enrollment.
8. No opportunistic infections in the past year.

   For less-well-controlled PLWH
9. PLWH with a CD4+ T-cell count of ≥ 200 and < 350 cells/μL at screening or viral load of 1,000 to 10,000 copies/mL.
10. PLWH being managed on a stable/unchanged (ART) regimen for at least 1 month prior to enrollment.

Exclusion Criteria:

1. Laboratory-confirmed SARS-CoV-2 infection (PCR+ within 5 days prior to first study vaccination with results available before randomization) or positive anti-S protein antibody to SARS-CoV-2 at screening.
2. Previous receipt of any investigational or authorized/approved vaccine, prophylactic or therapeutic agent for the prevention or treatment of COVID-19.
3. Participation in research involving receipt of an investigational product (drug/biologic/device) within 90 days prior to the first study vaccination.
4. Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine within 30 days prior to first study vaccination.
5. Any known allergies to products contained in the investigational product.
6. Any history of anaphylaxis to any prior vaccine.
7. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy.
8. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to first study vaccination.
9. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to first study vaccination.
10. Active cancer (malignancy) on therapy within 3 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
11. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.
12. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the first study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
13. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the trial vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
14. Study team member or immediate family member of any study team member (inclusive of Sponsor, Contract Research Organization, and study site personnel involved in the conduct or planning of the study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Number of PLWH with unsolicited adverse events (AEs) | Day 84
  Number of PLWH with unsolicited AEs stratified by level of control of HIV infection.
Number of HIV-Negative participants with unsolicited AEs | Day 84
  Number of HIV-Negative participants with unsolicited AEs.
Number of PLWH with unsolicited AEs | Day 120
  Number of PLWH with unsolicited AEs stratified by level of control of HIV infection.
Number of PLWH with unsolicited AEs | Day 180
  Number of PLWH with unsolicited AEs stratified by level of control of HIV infection.
Number of HIV-Negative participants with unsolicited AEs | Day 120
  Number of HIV-Negative participants with unsolicited AEs.
Number of HIV-Negative participants with unsolicited AEs | Day 180
  Number of HIV-Negative participants with unsolicited AEs.
Number of PLWH with solicited systemic AEs | Day 0
  Number of PLWH with solicited systemic AEs for 7 days following each vaccination stratified by baseline severity of disease as determined by the level of control of HIV infection into well-controlled and less-well-controlled treatment groups.
Number of PLWH with solicited systemic AEs | Day 21
  Number of PLWH with solicited systemic AEs for 7 days following each vaccination stratified by baseline severity of disease as determined by the level of control of HIV infection into well-controlled and less-well-controlled treatment groups.
Number of PLWH with solicited systemic AEs | Day 70
  Number of PLWH with solicited systemic AEs for 7 days following each vaccination stratified by baseline severity of disease as determined by the level of control of HIV infection into well-controlled and less-well-controlled treatment groups.
Number of HIV-Negative participants with solicited systemic AEs | Day 0
  Number of HIV-Negative participants with solicited systemic AEs for 7 days following each vaccination.
Number of HIV-Negative participants with solicited systemic AEs | Day 21
  Number of HIV-Negative participants with solicited systemic AEs for 7 days following each vaccination.
Number of HIV-Negative participants with solicited systemic AEs | Day 70
  Number of HIV-Negative participants with solicited systemic AEs for 7 days following each vaccination.
Number of PLWH with solicited local AEs | Day 0
  Number of PLWH with solicited local AEs for 7 days following each vaccination stratified by baseline severity of disease as determined by the level of control of HIV infection into well-controlled and less-well-controlled treatment groups.
Number of PLWH with solicited local AEs | Day 21
  Number of PLWH with solicited local AEs for 7 days following each vaccination stratified by baseline severity of disease as determined by the level of control of HIV infection into well-controlled and less-well-controlled treatment groups.
Number of PLWH with solicited local AEs | Day 70
  Number of PLWH with solicited local AEs for 7 days following each vaccination stratified by baseline severity of disease as determined by the level of control of HIV infection into well-controlled and less-well-controlled treatment groups.
Number of HIV-Negative participants with solicited local AEs | Day 0
  Number of HIV-Negative participants with solicited local AEs for 7 days following each vaccination.
Number of HIV-Negative participants with solicited local AEs | Day 21
  Number of HIV-Negative participants with solicited local AEs for 7 days following each vaccination.
Number of HIV-Negative participants with solicited local AEs | Day 70
  Number of HIV-Negative participants with solicited local AEs for 7 days following each vaccination.
Serum Immunoglobulin (IgG) antibody levels expressed as geometric mean enzyme-linked immunosorbent assay units (GMEU) | Day 21
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as GMEUs in PLWH stratified by level of control of HIV infection.
Serum Immunoglobulin (IgG) antibody levels expressed as geometric mean enzyme-linked immunosorbent assay units (GMEU) | Day 35
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as GMEUs in PLWH stratified by level of control of HIV infection.
Serum Immunoglobulin (IgG) antibody levels expressed as geometric mean enzyme-linked immunosorbent assay units (GMEU) | Day 70
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as GMEUs in PLWH stratified by level of control of HIV infection.
Serum Immunoglobulin (IgG) antibody levels expressed as geometric mean enzyme-linked immunosorbent assay units (GMEU) | Day 84
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as GMEUs in PLWH stratified by level of control of HIV infection.
Serum IgG antibody levels expressed as geometric mean fold rise (GMFR) | Day 21
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as GMFRs in PLWH stratified by level of control of HIV infection.
Serum IgG antibody levels expressed as geometric mean fold rise (GMFR) | Day 35
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as GMFRs in PLWH stratified by level of control of HIV infection.
Serum IgG antibody levels expressed as geometric mean fold rise (GMFR) | Day 70
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as GMFRs in PLWH stratified by level of control of HIV infection.
Serum IgG antibody levels expressed as geometric mean fold rise (GMFR) | Day 84
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as GMFRs in PLWH stratified by level of control of HIV infection.
Serum IgG antibody levels expressed as seroconversion rate (SCR) | Day 21
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as SCRs in PLWH stratified by level of control of HIV infection.
Serum IgG antibody levels expressed as seroconversion rate (SCR) | Day 35
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as SCRs in PLWH stratified by level of control of HIV infection.
Serum IgG antibody levels expressed as seroconversion rate (SCR) | Day 70
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as SCRs in PLWH stratified by level of control of HIV infection.
Serum IgG antibody levels expressed as seroconversion rate (SCR) | Day 84
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein antigen expressed as SCRs in PLWH stratified by level of control of HIV infection.
Human angiotensin-converting enzyme 2 (hACE2) receptor binding inhibition assay expressed as geometric mean titer (GMT) | Day 21
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as GMT in PLWH stratified by level of control of HIV infection.
Human angiotensin-converting enzyme 2 (hACE2) receptor binding inhibition assay expressed as geometric mean titer (GMT) | Day 35
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as GMT in PLWH stratified by level of control of HIV infection.
Human angiotensin-converting enzyme 2 (hACE2) receptor binding inhibition assay expressed as geometric mean titer (GMT) | Day 70
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as GMT in PLWH stratified by level of control of HIV infection.
Human angiotensin-converting enzyme 2 (hACE2) receptor binding inhibition assay expressed as geometric mean titer (GMT) | Day 84
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as GMT in PLWH stratified by level of control of HIV infection.
hACE2 receptor binding inhibition assay expressed as GMFR | Day 21
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as GMFR in PLWH stratified by level of control of HIV infection.
hACE2 receptor binding inhibition assay expressed as GMFR | Day 35
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as GMFR in PLWH stratified by level of control of HIV infection.
hACE2 receptor binding inhibition assay expressed as GMFR | Day 70
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as GMFR in PLWH stratified by level of control of HIV infection.
hACE2 receptor binding inhibition assay expressed as GMFR | Day 84
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as GMFR in PLWH stratified by level of control of HIV infection.
hACE2 receptor binding inhibition assay expressed as SCR | Day 21
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as SCR in PLWH stratified by level of control of HIV infection.
hACE2 receptor binding inhibition assay expressed as SCR | Day 35
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as SCR in PLWH stratified by level of control of HIV infection.
hACE2 receptor binding inhibition assay expressed as SCR | Day 70
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as SCR in PLWH stratified by level of control of HIV infection.
hACE2 receptor binding inhibition assay expressed as SCR | Day 84
  Epitope-specific immune responses assayed with the SARS-CoV-2 rS protein receptor-binding domain measured by serum titers in an hACE2 receptor binding inhibition assay expressed as SCR in PLWH stratified by level of control of HIV infection.
Neutralizing antibody activity expressed as GMT | Day 35
  Titers of neutralizing antibody to the prototype virus expressed as GMT in PLWH stratified by level of control of HIV infection.
Neutralizing antibody activity expressed as GMT | Day 84
  Titers of neutralizing antibody to the prototype virus expressed as GMT in PLWH stratified by level of control of HIV infection.
Neutralizing antibody activity expressed as SCR | Day 35
  Titers of neutralizing antibody to the prototype virus expressed as SCR in PLWH stratified by level of control of HIV infection.
Neutralizing antibody activity expressed as SCR | Day 84
  Titers of neutralizing antibody to the prototype virus expressed as SCR in PLWH stratified by level of control of HIV infection.
Neutralizing antibody activity expressed as GMFR | Day 35
  Titers of neutralizing antibodies to the prototype virus expressed as GMFR in PLWH stratified by level of control of HIV infection.
Neutralizing antibody activity expressed as GMFR | Day 84
  Titers of neutralizing antibodies to the prototype virus expressed as GMFR in PLWH stratified by level of control of HIV infection.

SECONDARY OUTCOMES:
Serum IgG antibody levels expressed as GMEU | Day 21
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as GMEUs in HIV-negative participants.
Serum IgG antibody levels expressed as GMEU | Day 35
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as GMEUs in HIV-negative participants.
Serum IgG antibody levels expressed as GMEU | Day 70
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as GMEUs in HIV-negative participants.
Serum IgG antibody levels expressed as GMEU | Day 84
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as GMEUs in HIV-negative participants.
Serum IgG antibody levels expressed as GMFR | Day 21
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as GMFR in HIV-negative participants.
Serum IgG antibody levels expressed as GMFR | Day 35
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as GMFR in HIV-negative participants.
Serum IgG antibody levels expressed as GMFR | Day 70
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as GMFR in HIV-negative participants.
Serum IgG antibody levels expressed as GMFR | Day 84
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as GMFR in HIV-negative participants.
Serum IgG antibody levels expressed as SCR | Day 21
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as SCR in HIV-negative participants.
Serum IgG antibody levels expressed as SCR | Day 35
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as SCR in HIV-negative participants.
Serum IgG antibody levels expressed as SCR | Day 70
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as SCR in HIV-negative participants.
Serum IgG antibody levels expressed as SCR | Day 84
  Serum IgG antibody levels assayed with the SARS-CoV-2 rS protein expressed as SCR in HIV-negative participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (7):
- South Africa (7):
  - KwaPhila Health Solutions (Enhancing Care), Westridge, Durban
  - Josha Research, Bloemfontein, Free State
  - The Aurum Institute Pretoria Clinical Research Services, Pretoria, Gauteng
  - Wits Vaccines & Infectious Diseases Analytics (VIDA) Research Unit, Diepkloof, Johannesburg
  - Wits RHI Shandukani Research Centre, Hillbrow, Johannesburg
  - MERC Research (Pty) Ltd - Middelburg, Middelburg, Mpumalanga
  - Madibeng Centre for Research, Brits, North West